CLINICAL TRIAL: NCT02486185
Title: Evaluation of the SARC-F Questionnaire, a New Screening Tool for Sarcopenia in People 65-year Old and Older in the Community
Brief Title: SARCORSICA: SARC-F Questionnaire as a Screening Tool for Age-related Sarcopenia
Acronym: SARCORSICA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-PP-19
Record Dates: First submitted 2015-04-01; First posted 2015-07-01 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SARC-F (Other): screening test for sarcopenia being studied, the SARC-F
  Interventions: Other: SCREENING TEST

INTERVENTIONS:
Other: SCREENING TEST — * Skeletal muscle mass, which will be estimated by calculating values for the mid-arm muscle circumference (MAMC) from brachial perimeter (BP) and triceps skinfold thickness (TSF).
  * Muscle force will be measured using a hydraulic dynamometer
  * Physical performance will be estimated from the subject's Gait speed using a 4 meter gait test (Gait speed 4-m)

SUMMARY:
Background to the research: Sarcopenia is a geriatric syndrome defined by progressive generalised loss of skeletal muscle, mass, force and function.

Problem statement and objectives: To validate a simple, reproducible, screening tool, which is easy to use in the general practitioner's surgery is one of the challenges of the future.

The primary objective is to assess the sensitivity and specificity of the study screening test, the SARC-F, at a predetermined threshold of >= 4. A total score of >=4 is associated with poor physical performance and is also predictive of the clinical diagnosis of the disease. The secondary objectives are to assess the prevalence of sarcopenia in the study population, to carry out a subgroup analysis of statistical performance for the five questions tested by the SARC-F, to identify the main risk factors associated with the disease and to propose an algorithm, positioning the SARC-F at the heart of a systematic screening process for the disease.

Materials and methods: This is a diagnostic, cross-sectional study with a descriptive and analytical epidemiological component to analyse the secondary endpoints. It will be carried out in usual care over a period of 6 months in a homogeneous population of 65-year-old and older patients from the community consulting in primary care. The subjects will undergo the screening test (SARC-F questionnaire) and then the reference clinical assessment (gold standard) in succession.

Expected results: To demonstrate the statistical tests that the SARC-F questionnaire is a simple tool, appropriate for early screening of sarcopenia in primary care.

DETAILED DESCRIPTION:
Background to the research: Sarcopenia is a multifactorial geriatric syndrome with a prevalence ranging between 1 and 29% depending on age. It is defined by progressive, generalised loss of skeletal muscle, mass, force and function.

Problem statement and objectives: To confirm a simple, reproducible, screening tool, which is easy to use in the general practitioner's surgery is one of the challenges of the future.

The primary objective is to assess the sensitivity and specificity of the study screening test, the SARC-F, at a predetermined threshold of >=4 and to change this threshold using a ROC curve to attempt to increase its sensitivity. This questionnaire has been shown to provide low sensitivity (4%-10%) but high specificity (94%-99%) in the study carried out by Woo and co-workers on an analysis of statistical performance of the questionnaire, stratified by sex. A total score of >= 4 is associated with poor physical performance and is also predictive of the clinical diagnosis of the disease. The test will be assessed compared to the clinical diagnosis of the disease using international criteria recognised by EWGSOP, which defines sarcopenia as a reduction in muscle mass, associated with a reduction in muscle force and/or reduced physical performance by the subject. The secondary objectives are to assess the prevalence of sarcopenia in the study population, to carry out a sub-group analysis of the statistical performance of the five questions tested by the SARC-F and to identify the main risk factors associated with the disease and finally to propose an algorithm positioning the SARC-F at the heart of a systematic screening process for the disease.

Materials and Methods: This is a diagnostic, cross-sectional study with a descriptive and analytical epidemiological component to analyse the secondary end points. It will be carried out in usual care over a period of 6 months. The study will be conducted in Southern Corsica in a homogeneous population of 65 year old and older patients from the community, consulting in primary care. The number of subjects required is calculated for a disease prevalence set at 15%, a 95% specificity for the screening test with a minimum acceptable confidence interval of 80%. A total of 366 patients will therefore need to be included. The subjects will undergo the screening test (SARC-F questionnaire) and then the reference clinical assessment (gold standard) in succession). Muscle force will be assessed using a dynamometer, physical performance by a 4-metre gait test and brachial muscle circumference (BMC) will be calculated from two simple anthropometric measurements, the tricipital skin fold thickness (TS) and the brachial perimeter (BP).

Expected results: To demonstrate the statistical tests that the SARC-F questionnaire is a simple tool, appropriate for early screening of sarcopenia in primary care; to define a new optimal threshold achieving greater sensitivity, to make practitioners aware of screening for sarcopenia, to improve its prevention and to promote its management as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* Men or women who are 65-year old or older consulting a general practitioner, regardless of initial reason for the consultation.
* Patients agreeing to take part in the study after clear, true and appropriate information has been provided, giving their signed consent and having been given by hand a patient information sheet.

exclusion criteria:

* Patients with cognitive disorders suffering from major incapacity making understanding the study or signing the informed consent impossible.
* Patients not affiliated to a Social Security system.
* Patients suffering from acute functional problems interfering with the tests being performed (incapacity, malformation of the arm, plaster or splint).
* Patients institutionalised in nursing homes or subacute care
* Patients who use a technical aid for walking, unless this aid is a walking stick
* Patients not being followed up in a general practitioner's surgery (absence of information required to carry out the analytical part)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 366 (Actual)
Dates: Start 2014-11-16 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
questionnaire SARC-F | thirty minutes

SECONDARY OUTCOMES:
number of participant | thirty minutes

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane M SCHNEIDER, Principal Investigator — schneider.s@chu-nice.fr
Locations (2):
- France (2):
  - Cabinet de Médecine Générale, Cozzano, Corsica
  - Cabinet de médecine générale, Peri, Corsica